CLINICAL TRIAL: NCT04709432
Title: Extracorporeal Membrane Oxygenation (ECMO) Treatment of Children in Mainland China in the Past 10 Years
Brief Title: ECMO Treatment of Children in China in the Past 10 Years
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-06
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Extracorporeal Membrane Oxygenation; Child, Only
Keywords: Extracorporeal membrane oxygenation; children; complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO group: children supported by ECMO in the past 10 years
  Interventions: Procedure: ECMO

INTERVENTIONS:
Procedure: ECMO — ECMO is a form of Extracorporeal Life Support (ECLS) to support either the pulmonary, or both the pulmonary and cardiac systems.

SUMMARY:
It is a cross-sectional study to summarize the extracorporeal membrane oxygenation （ECMO）treatment in children in China.

DETAILED DESCRIPTION:
ECMO treatment in children is still in its infancy in China, and it has made considerable progress in recent years. In order to further understand the development of ECMO treatment in critically ill children, the investigator conduct this cross-sectional research through questionnaires. The investigator collect general information of the hospital and ECMO equipment, etiology, compilation, and mode of ECMO.

ELIGIBILITY:
Inclusion Criteria:

* age of 1d to 18 years old;
* children supported by ECMO in mainland China in the past 10 years

Exclusion Criteria:

* none

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children supported by ECMO in mainland China in the past years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
survival rate | from admission to discharge （about 10days）
  survival rate after discharge

SECONDARY OUTCOMES:
time of running ECMO | from admission to discharge（about 10days）
  the total time of running ECMO
cost of ECMO treatment | from admission to discharge （about 10days）
  the total cost of ECMO treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lu Guoping, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China